CLINICAL TRIAL: NCT03647488
Title: Phase II Multicenter Randomized Two-arm Study of Capmatinib and Spartalizumab Combination Therapy vs Docetaxel in Pretreated Adult Patients With EGFR Wild-type ALK Rearrangement Negative Advanced/Metastatic Non-small Cell Lung Cancer
Brief Title: Study of Capmatinib and Spartalizumab Combination Therapy vs Docetaxel in Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280D2201; 2018-001420-19 (EudraCT Number)
Record Dates: First submitted 2018-08-20; First posted 2018-08-27 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small-cell lung carcinoma; Non-small-cell lung cancer; NSCLC; epidermal growth factor receptor wild type; EGFRwt; Anaplastic lymphoma kinase negative; ALK-; INC280; capmatinib and spartalizumab; combination therapy; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib; spartalizumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Run-in part was single group. Randomized part (parallel design) was not opened.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Run-in part: capmatinib + spartalizumab (Experimental): Participants (enrolled in the run-in part) were treated with capmatinib 400 mg twice daily (BID) and spartalizumab 400 mg intravenously (i.v.) once every 28 days
  Interventions: Drug: Capmatinib; Drug: Spartalizumab
- Randomized part: capmatinib+spartalizumab (Experimental): Participants (enrolled in the randomized part) treated with capmatinib 400 mg twice daily (BID) and spartalizumab 400 mg intravenously (i.v.) once every 28 days
  Interventions: Drug: Capmatinib; Drug: Spartalizumab
- Randomized part: docetaxel (Active Comparator): Participants (enrolled in the randomized part) treated with docetaxel 75mg/m2 i.v. following local guidelines as per standard of care and product labels once every 21 days
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Capmatinib — Capmatinib 400 mg (tablets) orally taken twice daily
  Other Names: INC280
  Arms: Randomized part: capmatinib+spartalizumab; Run-in part: capmatinib + spartalizumab
Drug: Spartalizumab — Spartalizumab 400 mg via intravenous infusion once every 28 days
  Other Names: PDR001
  Arms: Randomized part: capmatinib+spartalizumab; Run-in part: capmatinib + spartalizumab
Drug: Docetaxel — Docetaxel 75mg/m2 i.v. following local guidelines as per standard of care and product labels once every 21 days
  Arms: Randomized part: docetaxel

SUMMARY:
The purpose of this trial was to evaluate the safety and efficacy of capmatinib in combination with spartalizumab in adult participants with epidermal growth factor receptor (EGFR) wild type (for exon 19 deletions and exon 21 L858R substitution mutations), anaplastic lymphoma kinase (ALK) rearrangement negative in locally advanced (stage IIIB, not eligible for definitive chemo-radiation) or metastatic (stage IV) Non-small cell lung cancer (NSCLC) after failure of platinum doublet and checkpoint inhibitor treatment.

DETAILED DESCRIPTION:
This was a two-part prospectively designed, multicenter, open-label, randomized phase II study.

Part 1: Run-in. Prior to the randomized part of the study, a run-in to assess the safety and tolerability as well as preliminary efficacy of the capmatinib and spartalizumab combination was conducted. Participants were treated with capmatinib 400 mg twice daily (BID) and spartalizumab 400 mg intravenously (i.v.) once every 28 days. A review was planned to take place after all participants had at least 24 weeks of follow-up. The decision to expand the study to the randomized part was to be based on the safety, tolerability, and preliminary efficacy of the capmatinib and spartalizumab combination.

Part 2: Randomized. Subjects were planned to be randomized to one of the following arms in a 2:1 ratio: 1) combination of capmatinib 400 mg BID and spartalizumab 400 mg i.v. once every 28 days; 2) docetaxel 75 mg/m2 i.v. following local guidelines as per standard of care and product labels. Based on the results obtained in the run-in part of the study, the randomized part was not opened.

For the run-in part of the study, the treatment period began on Cycle 1 Day 1 and continued in 28-day cycles until disease progression, unacceptable toxicity, withdrawal of informed consent, pregnancy, lost to follow-up, or death irrespective of start of new anti-neoplastic therapy. After treatment discontinuation, all subjects were followed for safety evaluations during the safety follow-up period, and the subject's status was collected every 8 weeks as part of the survival follow-up

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced/metastatic (stage IIIB/IV), EGFR wild-type, ALK rearrangement negative, non-small cell lung cancer
* Subject had demonstrated progression following one prior platinum doublet and one prior PD-(L)1 checkpoint inhibitor (either alone or in combination, the most recent treatment regimen must have contained a PD-(L)1 checkpoint inhibitor)
* Subjects must be candidates for single agent docetaxel
* Subjects must have at least one lesion evaluable by RECIST 1.1

Exclusion Criteria:

* Prior treatment with a MET inhibitor or HGF (Hepatocyte growth factor) targeting therapy
* Any untreated central nervous system (CNS) lesion
* Use of any live vaccines against infectious diseases within 12 weeks of initiation of study treatment.

Other protocol-defined inclusion/exclusion criteria might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Highlands Oncology Group, Fayetteville, Arkansas, United States
- Novartis Investigative Site, Leuven, Belgium
- France (2):
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille Cédex
- Novartis Investigative Site, Cologne, Germany
- Novartis Investigative Site, Tel Aviv, Israel
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Plain language trial summaries are available on this link — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=883

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on preliminary results of run-in part, the decision was not to open randomized part of the study. Therefore, no participants were enrolled in randomized part.
Groups:
- Randomized Part: Capmatinib + Spartalizumab: Participants (enrolled in the randomized part) treated with capmatinib 400 mg twice daily (BID) and spartalizumab 400 mg intravenously (i.v.) once every 28 days
Period: Overall Study
Arm/Group | Run-in Part: Capmatinib + Spartalizumab | Randomized Part: Capmatinib + Spartalizumab | Randomized Part: Docetaxel
Started | 18 | 0 (Randomized part was not opened) | 0 (Randomized part was not opened)
Completed | 0 | 0 | 0
Not Completed | 18 | 0 | 0
Not completed — Progressive disease | 10 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Clinical progression | 2 | 0 | 0
Not completed — Participant refused to take investigational product | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Based on preliminary results of run-in part, randomized part was not opened. Therefore, no participants were enrolled in the randomized part of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-in Part: Capmatinib + Spartalizumab | Randomized Part: Capmatinib + Spartalizumab | Randomized Part: Docetaxel | Total
Number analyzed (Participants) | 18 | 0 | 0 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (10.52) |  |  | 61.2 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 0 | 7
  Male | 11 | 0 | 0 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 0 | 0 | 17
  Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Run-in Part: Percentage of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as an adverse event or abnormal laboratory value assessed as unrelated to disease progression, inter-current illness, or concomitant medications that met certain criteria as defined in the protocol.
Time Frame: From the day of the first dose of study medication up to 56 days
Population: All participants from the Safety Set in the run-in who experienced DLT during the first 8 weeks of dosing or met the minimum exposure criterion (subject received at least 1 infusion of spartalizumab and took at least 50% of the planned dose of capmatinib within the first 8 weeks of treatment) and had sufficient safety evaluations (subjects were observed for ≥56 days following the first dose, and are considered to have enough safety data to conclude that a DLT did not occur).
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Participants | 1

2. Primary Outcome: Run-in Part: Percentage of Participants With Adverse Events (AEs)
Description: Percentage of participants with AEs, including changes from baseline in vital signs and laboratory results qualifying and reported as AEs.
  AEs were assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0: Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: Death
Time Frame: From the day of the first dose of study medication to 150 days after the last dose of spartalizumab, or 30 days after the last dose of capmatinib (whichever is later) up to maximum duration of approximately 1.7 years
Population: All participants in the run-in who received at least one dose of study treatment (i.e. at least one dose of spartalizumab [including incomplete infusion] or of capmatinib).
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Participants
  AEs- All grades | 18
  AEs- Grade ≥3 | 11
  Treatment-related AEs- All grades | 14
  Treatment related AEs- Grade ≥3 | 1
  Serious AEs (SAEs)- All grades | 10
  SAEs- Grade ≥3 | 7
  Treatment-related SAEs- All grades | 3
  Treatment-related SAEs- Grade ≥3 | 0
  Fatal SAEs- All grades | 1
  Fatal SAEs- Grade ≥3 | 1
  AEs leading to discontinuation- All grades | 5
  AEs leading to discontinuation- Grade ≥3 | 3
  Treatment-related AEs leading to discontinuation- All grades | 3
  Treatment-related AEs leading to discontinuation- Grade ≥3 | 1
  AEs leading to dose adjustment/interruption- All grades | 9
  AEs leading to dose adjustment/interruption- Grade ≥3 | 5
  AEs requiring additional therapy- All grades | 16
  AEs requiring additional therapy- Grade ≥3 | 8

3. Primary Outcome: Run-in Part: Percentage of Participants With at Least One Dose Reduction.
Description: Percentage of participants with at least one dose reduction. Dose reductions were only allowed for capmatinib
Time Frame: From the day of the first dose of study medication to end of treatment, assessed up to maximum duration of 68 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Participants | 6

4. Primary Outcome: Run-in Part: Percentage of Participants With at Least One Dose Interruption
Description: Percentage of participants with at least one dose interruption. Dose interruptions were allowed for capmatinib and spartalizumab.
Time Frame: From the day of the first dose of study medication to end of treatment, assessed up to maximum duration of 68 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Participants
  Capmatinib | 8
  Spartalizumab | 3

5. Primary Outcome: Run-in Part: Relative Dose Intensity Received by Participants
Description: The relative dose intensity of capmatinib and spartalizumab is computed as the ratio of dose intensity and planned dose intensity, multiplied by 100.
Time Frame: From the day of the first dose of study medication to end of treatment, assessed up to maximum duration of 68 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage of dose received
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Percentage of dose received
  Capmatinib | 99.6 [27.8 to 100.0]
  Spartalizumab | 100.0 [75.0 to 133.3]

6. Primary Outcome: Randomized Part: Overall Survival (OS)
Description: OS is defined as the time from date of start of treatment to date of death due to any cause. If a participant was not known to have died, survival was censored at the date of last known date patient alive.
  Results are not available because randomized part never started.
Time Frame: From start of treatment to death due to any cause, assessed until the end of the study (up to a planned duration of 18 months)
Population: Data was not collected as no participants were enrolled in randomized part.
Arm/Group | Randomized Part: Capmatinib + Spartalizumab | Randomized Part: Docetaxel
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Objective Response Rate (ORR) Based on RECIST 1.1 and as Per Investigator Assessment
Description: ORR is defined as the percentage of subjects with best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and as per investigator assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  ORR results for randomized part are not available because randomized part never started.
Time Frame: From start of treatment until end of treatment, assessed up to 68 weeks (run-in part)
Population: All participants in the run-in who received at least one dose of any component of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Percentage of participants | 0 [0.0 to 18.5]

8. Secondary Outcome: Disease Control Rate (DCR) Based on RECIST 1.1 and as Per Investigator Assessment
Description: DCR is defined as the percentage of subjects with best overall response of CR or PR or stable disease based on RECIST 1.1 and as per investigator assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  Stable disease: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
  DCR results for randomized part are not available because randomized part never started.
Time Frame: From start of treatment until end of treatment, assessed up to 68 weeks (run-in part)
Population: All participants in the run-in who received at least one dose of any component of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Percentage of participants | 27.8 [9.7 to 53.5]

9. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented radiological progression or death due to any cause. For participants who had not progressed or died at the analysis cut-off date, PFS was censored at the date of the last adequate tumor evaluation date. An adequate tumour assessment is a tumour assessment with an overall response other than unknown.
  Progression is defined using RECIST 1.1 and as per investigator assessment as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  PFS results for randomized part are not available because randomized part never started.
Time Frame: From start of treatment until the first documented radiological progression or death, whichever comes first, assessed up to 68 weeks (run-in part)
Population: All participants in the run-in who received at least one dose of any component of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Months | 1.9 [1.7 to 3.6]

10. Secondary Outcome: Time to Response (TTR) Based on RECIST 1.1 and as Per Investigator Assessment
Description: TTR is defined as the time from the date of start of treatment to the first documented response of either CR or PR, which must be subsequently confirmed. TTR was evaluated according to RECIST 1.1 and as per investigator assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  For run-in part, TTR results are not available because there were no participants achieving response (CR or PR) For randomized part , TTR results are not available because randomized part never started.
Time Frame: From start of treatment to the first documented response of either complete response or partial response, assessed up to 68 weeks (run-in part)
Population: No data available as no participants had event
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Duration of Response (DOR) Based on RECIST 1.1 and as Per Investigator Assessment
Description: DOR is the time between the date of first documented response(CR or PR) and the date of first documented progression or death due to underlying cancer based on RECIST1.1 and as per investigator assessment. If progression or death has not occurred, the subject is censored at the date of last adequate tumor assessment. CR: Disappearance of all non-nodal target lesions and any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Progression: at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. The sum must also demonstrate an absolute increase of at least 5 mm. Results are not available because there were no participants achieving response in the run-in part and randomized part never started
Time Frame: From first documented response (CR or PR) to first documented progression or death, whichever came first, assessed up to 68 weeks (run-in part)
Population: No data available as no participants had event
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 0

12. Secondary Outcome: AUClast of Capmatinib
Description: AUClast is the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration. AUClast was calculated using non-compartmental methods.
Time Frame: Cycle 3 day 1 at predose, 0.5 hours (h), 1h, 2h, 4h and 8h postdose. Each Cycle is 28 days
Population: The capmatinib pharmacokinetic (PK) analysis set included all participants in the run-in phase who provided at least one evaluable capmatinib PK concentration. Only those participants with data available for this endpoint at specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 8
nanogram*hour/milliliter (ng*hr/mL) | 11500 (47.3)

13. Secondary Outcome: AUCtau of Capmatinib
Description: AUCtau is the area under the plasma concentration-time curve from time zero to the end of the dosing interval Tau. AUCtau was calculated using non-compartmental methods.
Time Frame: Cycle 3 day 1 at predose, 0.5 hours (h), 1h, 2h, 4h and 8h postdose. Each Cycle is 28 days
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 5
nanogram*hour/milliliter (ng*hr/mL) | 12800 (48.5)

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Capmatinib
Description: The maximum (peak) observed plasma concentration after single dose administration. Cmax was calculated using non-compartmental methods.
Time Frame: Cycle 3 day 1 at predose, 0.5 hours (h), 1h, 2h, 4h and 8h postdose. Each Cycle is 28 days
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 8
nanogram/milliliter (ng/mL) | 3260 (44.6)

15. Secondary Outcome: Time to Reach Maximum (Tmax) Plasma Concentration of Capmatinib
Description: Tmax is the time to reach maximum (peak) plasma concentration of capmatinib after single dose administration (time). Tmax was calculated using non-compartmental methods.
Time Frame: Cycle 3 day 1 at predose, 0.5 hours (h), 1h, 2h, 4h and 8h postdose. Each Cycle is 28 days
Population: as for outcome 12
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 8
hour (h) | 1.42 [0.983 to 2.00]

16. Secondary Outcome: AUClast of Spartlizumab
Description: as for outcome 12
Time Frame: CCycle 3 day 1 at predose and 1 hour postdose (up to 1.53 hours postdose), cycle 3 day 4 (=72 hours postdose), cycle 3 day 8 (=168 hours postdose) and cycle 3 day 15 (=336 hours postdose). Each Cycle is 28 days
Population: The spartlizumab pharmacokinetic (PK) analysis set included all participants in the run-in phase who provided at least one evaluable spartlizumab PK concentration. Only those participants with data available for this endpoint at specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter (μg*day/mL)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 7
microgram*day/milliliter (μg*day/mL) | 1720 (64.5)

17. Secondary Outcome: AUCtau of Spartlizumab
Description: as for outcome 13
Time Frame: Cycle 3 day 1 at predose and 1 hour postdose (up to 1.53 hours postdose), cycle 3 day 4 (=72 hours postdose), cycle 3 day 8 (=168 hours postdose) and cycle 3 day 15 (=336 hours postdose). Each Cycle is 28 days
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter (μg*day/mL)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 7
microgram*day/milliliter (μg*day/mL) | 2110 (35.1)

18. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Spartlizumab
Description: as for outcome 14
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 8
microgram/milliliter (μg/mL) | 138 (23.2)

19. Secondary Outcome: Time to Reach Maximum (Tmax) Plasma Concentration of Spartlizumab
Description: Tmax is the time to reach maximum (peak) plasma concentration of spartlizumab after single dose administration (time). Tmax was calculated using non-compartmental methods.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 8
hour (h) | 1.13 [1.00 to 1.53]

20. Secondary Outcome: Spartalizumab Antidrug Antibodies (ADA) Prevalence at Baseline
Description: ADA prevalence at baseline was calculated as the proportion of participants who had an ADA positive result at baseline
Time Frame: Cycle 1 Day 1 at predose. Each Cycle is 28 days
Population: immunogenicity (IG) prevalence set includes all subjects in the Full analysis set with a determinant baseline IG sample or at least one determinant post-baseline sample.
  Determinant sample: sample that is neither ADA-inconclusive nor unevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 17
Participants | 3

21. Secondary Outcome: Spartalizumab ADA Incidence On-treatment
Description: ADA incidence on treatment was calculated as the proportion of participants who were treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: Predose at Cycle (C)1 Day (D)1, C2D1, C3D1, C4D1, C6D1, C8D1, C10D1, C12D1, thereafter every 6 cycles until discontinuation, and end of treatment (EOT), 30-day and 150-day after EOT
Population: The IG incidence set includes all subjects in the IG prevalence set with a determinant baseline IG sample and at least one determinant post-baseline IG sample.
  Determinant sample: sample that is neither ADA-inconclusive nor unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 14
Participants | 3

22. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths due to any cause were collected from first dose of study medication to 150 days after the last dose of spartalizumab, or 30 days after the last dose of capmatinib, whichever is later, up to a maximum duration of approximately 1.7 years.
  Total deaths were collected from first dose of study treatment until end of post-treatment efficacy or survival follow, up to maximum duration of approximately 1.7 years
Time Frame: On-treatment deaths: up to approximately 1.7 years. All deaths: up to approximately 1.7 years
Population: Safety Set consisted of all participants who received at least one dose of study treatment, i.e. at least one dose of spartalizumab [including incomplete infusion] or of capmatinib.
Measure: Number; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
Number analyzed (Participants) | 18
Participants
  Total Deaths | 12
  Deaths on-treatment | 5

ADVERSE EVENTS:
Time Frame: On-treatment deaths due to any cause and adverse events were collected from first dose of study medication to 150 days after the last dose of spartalizumab, or 30 days after the last dose of capmatinib, whichever is later, up to a maximum duration of approximately 1.7 years.
Description: Any sign or symptom that occurs during the study treatment plus 150 days after the last dose of spartalizumab or 30 days after the last dose of capmatinib (on-treatment). Total number of deaths are captured in Outcome Measure 22 (post-hoc: all-cause mortality). Analysis performed on the safety set in the run-in part: all participants who received at least one dose of spartalizumab [including incomplete infusion] or of capmatinib. No safety data is available for part 2 because it was not opened.
Arm/Group | Run-in Part: Capmatinib + Spartalizumab
All-Cause Mortality (participants affected / at risk) | 5/18
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Part: Capmatinib + Spartalizumab (N=18)
Cardiac failure congestive (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Fatigue (General disorders) | 3
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Abdominal infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Part: Capmatinib + Spartalizumab (N=18)
Anaemia (Blood and lymphatic system disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Eyelid oedema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 4
Axillary pain (General disorders) | 1
Chest pain (General disorders) | 2
Fatigue (General disorders) | 4
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Herpes zoster (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 5
Blood magnesium decreased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
Creatinine renal clearance decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT03647488/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03647488/SAP_001.pdf